CLINICAL TRIAL: NCT02774993
Title: Doxycycline and the Modulation of Host Immunopathology in Human Pulmonary Tuberculosis: A Pilot Study
Brief Title: Doxycycline in Human Pulmonary Tuberculosis
Acronym: Doxy-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other); National University of Singapore (Other); A*Star (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Doxy_TB
Record Dates: First submitted 2016-03-11; First posted 2016-05-17 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2016-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Experimental): Doxycycline 100 mg twice daily with once daily anti-tuberculous treatment comprising of rifampicin 10 mg/kg, isoniazid 5 mg/kg, ethambutol 20 mg/kg, pyrazinamide 25 mg/kg and pyridoxine 10-50 mg per day according to managing physicians' discretion. These will be given daily for 14 days. Subsequently doxycycline will be ceased and patients are to continue with their standard anti-tuberculous treatment and duration according to their managing physician
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Placebo twice daily with once daily anti-tuberculous treatment comprising of rifampicin 10 mg/kg, isoniazid 5 mg/kg, ethambutol 20 mg/kg, pyrazinamide 25 mg/kg and pyridoxine 10-50 mg per day according to managing physicians' discretion. These will be given daily for 14 days. Subsequently placebo will be ceased and patients are to continue with their standard anti-tuberculous treatment and duration according to their managing physician
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Doxycycline
  Arms: Doxycycline
Drug: placebo
  Arms: Placebo

SUMMARY:
Pulmonary cavitation, a hallmark of tuberculosis (TB), is the site of high mycobacterial burden leading to disease transmission. The cause of tissue destruction leading to cavitation in TB is primarily due to the host inflammatory response. A matrix degrading phenotype develops in TB, in which the activity of host proteolytic enzymes, specifically matrix metalloproteinases (MMPs) is unopposed by their specific Tissue Inhibitors of Metalloproteinases (TIMPs), thus driving tissue destruction and cavitation in TB. This tissue destruction causes morbidity and mortality. MMP inhibition with doxycycline has shown to improve lung function in patients with chronic lung diseases but its use in TB is unclear.

We hypothesise that the MMP inhibitor doxycycline will reduce tissue destruction in human pulmonary tuberculosis.

Specific aims:

* To investigate the MMP and TIMP secretion and gene expression in M. tuberculosis (M.tb) - infected primary neutrophils and monocytes from healthy volunteers taking doxycycline.
* To investigate the intracellular signaling pathways modulated by doxycycline
* To investigate the effects doxycycline has on biological markers of tissue destruction in TB patients
* To assess the tolerability and side effects of doxycycline with concurrent standard TB therapy

DETAILED DESCRIPTION:
All TB patients are to keep to their standard anti-tuberculous treatment. A standardized questionnaire of symptoms, side-effects and weight shall be recorded. Induced sputum and plasma samples from all TB patients shall be analysed for MMPs and TIMPs before and after the administration of doxycycline for two weeks. In addition, neutrophils and mononuclear cells from TB patients and these shall be stimulated with live, virulent M. tuberculosis in a Biosafety Level 3 laboratory. The supernatants from these cells shall be analysed for MMPs and TIMPs.

Healthy volunteers shall be recruited and administered doxycycline for 2 weeks. Neutrophils and mononuclear cells will be isolated from blood prior to treatment, at weeks 2 and 8 and infected with M.tb. Cell culture supernatants and nucleic acids will be harvested. MMP and TIMP expression will be analysed using luminex array and real-time polymerase chain reaction. Intracellular signaling pathways will be examined with a human phospho-kinase array. Matrix destruction will be assessed using collagen quantitative fluorescent assays.

ELIGIBILITY:
Healthy Volunteers 10 volunteers will be recruited comprising 5 females and 5 males.

Inclusion criteria:

1. No known medical conditions
2. Aged 21 years to less than 70.

Exclusion criteria:

1. Unable to give informed consent
2. Prisoners
3. Pregnancy or nursing
4. On medication or oral contraceptives
5. Any concurrent illness, such as influenza

TB patients

Inclusion criteria: Patients should meet all criteria

1. Patients receiving ≤ 7 days of TB treatment or about to start standard combination TB treatment
2. Confirmed pulmonary TB with positive acid-fast bacilli smear and/or positive TB GeneXpert test and/or culture results
3. Chest radiograph demonstrating pulmonary involvement
4. Aged 21 years to less than 70

Exclusion criteria:

1. HIV co-infection
2. Previous pulmonary TB
3. Severe, pre-existing lung disease such as pulmonary fibrosis, bronchiectasis, Chronic obstructive pulmonary disease and lung cancer
4. Pregnant or breast feeding
5. Allergies to tetracyclines
6. Patients on retinoic acid, neuromuscular blocking agents and pimozide which may increase risk of drug toxicity
7. Autoimmune disease and/or on systemic immunosuppressants
8. Unable to provide informed consent
9. Haemoglobin < 8 g/dl
10. Creatinine 2 times upper limit of normal (ULN)
11. Alanine transaminase >3 times ULN
12. Use of any investigational or non-registered drug, vaccine or medical device other than the study drug within 182 days preceding dosing of study drug, or planned use during the study period
13. Enrolment in any other clinical trial involving a systemic drug or intervention involving the lung
14. Evidence of severe depression, schizophrenia or mania
15. Principal investigator assessment of lack of willingness to participate and comply with all requirements of the protocol, or identification of any factor felt to significantly increase the participant's risk of suffering an adverse outcome

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change of serum marker Procollagen III N-terminal peptide (PIIINP) from day 0 to day 14 in TB patients | Day 0 and Day 14

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | day 0 to day 56

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Miow QH, Vallejo AF, Wang Y, Hong JM, Bai C, Teo FS, Wang AD, Loh HR, Tan TZ, Ding Y, She HW, Gan SH, Paton NI, Lum J, Tay A, Chee CB, Tambyah PA, Polak ME, Wang YT, Singhal A, Elkington PT, Friedland JS, Ong CW. Doxycycline host-directed therapy in human pulmonary tuberculosis. J Clin Invest. 2021 Aug 2;131(15):e141895. doi: 10.1172/JCI141895. PMID 34128838